CLINICAL TRIAL: NCT05368233
Title: Impact of Abdominal Drains on the Efficacy of ERAS Pathway in the Perioperative Management of Peptic Perforation - A Randomized Control Trail (TUBELESS TRAIL)
Brief Title: Impact of Abdominal Drains on the ERAS Pathway in Peptic Perforation
Acronym: TUBELESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Tushar Subhadarshan Mishra, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG Thesis/2021-22/111
Record Dates: First submitted 2022-04-08; First posted 2022-05-10 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Perforated Peptic Ulcer; Fast Track Surgery; Perforated Bowel; Post-Op Complication; Emergencies
Keywords: ERAS; Emergency surgery; fast track surgery; perioperative care; Enhanced recovery after surgery
MeSH Terms: conditions — Peptic Ulcer Perforation; Intestinal Perforation; Postoperative Complications; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS protocol without the use of of abdominal drain in the perforated peptic ulcer patient (Experimental): Tracheal intubation. Short acting anesthetic agents,avoid opioid agents . Omental patch repair without placement of sub hepatic drain. Bilateral Transverse abdominis plane block/ Rectus sheath block immediately after surgery.
  Abdominal drain will not be placed Post operative nausea and vomiting prophylaxis. Encourage to mobilize out of bed after effect of general anesthesia has weaned off.
  Initiation of feeding-Oral sips on day 1, step up day 2 onward. Removal of nasogastric tube-immediately after surgery after aspirating the gastric content through nasogastric tube.
  Removal of urinary catheter-after weaning from the effect of general anesthesia.
  Avoid opioid analgesics.
  Interventions: Other: ERAS protocol
- ERAS protocol with the use of of abdominal drain in the perforated peptic ulcer patient (Active Comparator): Tracheal intubation. Short acting anesthetic agents, avoid opioid agents. Omental patch repair with placement of sub hepatic drain. Bilateral Transverse abdominis plane block/ Rectus sheath block immediately after surgery.
  Abdominal Drains will be placed and removed at anytime within 24 hrs and to not remove if the output is bilious or pus.
  Post operative nausea and vomiting prophylaxis. Encourage to mobilize out of bed after effect of general anesthesia has weaned off.
  Initiation of feeding-Oral sips on day 1, step up day 2 onward. Removal of nasogastric tube-immediately after surgery after aspirating the gastric content through nasogastric tube.
  Removal of urinary catheter-after weaning from the effect of general anesthesia.
  Placing Sub hepatic drain intraoperatively. Avoid opioid analgesics.
  Interventions: Other: ERAS protocol

INTERVENTIONS:
Other: ERAS protocol — ERAS protocol whch helps to optimise the length of hospital stay.
  Other Names: Fast track study

SUMMARY:
This study plans to assess the effect of placement of abdominal drains on the outcomes of ERAS (Enhanced recovery after surgery) protocol in the perioperative management of peptic perforation. In the study arm ERAS protocol will be implemented avoiding use of abdominal drain. In the control arm abdominal drains will be placed in the early post operative period while using the ERAS protocol. The effect of drains on duration of post operative stay and other return to physiological parameter like onset of ambulation, oral intake, passing flatus and feces etc. will be studied. The investigators hypothesize that the non-placement of abdominal drain postoperatively will not have worse outcomes than in cases where it is used postoperatively, in terms of length of hospital stay.

.

DETAILED DESCRIPTION:
ERAS is a an evidence based perioperative care pathways aiming reduction in the surgical stress. ERAS is a an evidence based perioperative care pathways aiming reduction in the surgical stress. Studies assessing the outcome of non usage to abdominal drains on the post-operative outcomes are scarce. This study aims to study the influence of abdominal drains on the post operative hospital stay and other functional outcomes.

Methods Patient with hollow viscus perforation to the emergency rooms and diagnosed to have peptic ulcer perforation intraoperatively will be included in the study. After omental patch repair and completion of operative procedure, patient will be randomized into drain group and no drain group based on the random allocation software.

Preoperative Early identification of physiological derangement and intervention. Early identification of physiological derangement and intervention. Early identification of physiological derangement and intervention. Early imaging , surgery and source control of sepsis. Risk assessment - PULP (Peptic Ulcers Perforation) score, Mannheim peritonitis index score, Boey score.

Intraoperatively Short acting anesthesia agents. warm normal saline lavage. Omental patch repair. Bilateral rectus sheath block. Bilateral rectus sheath block. Peritoneal fluid for culture and sensitivity. Mucosal edge / pinch biopsy to rule out any malignancy. Post operative nausea and vomiting (PONV) prophylaxis Balanced intravenous fluid administration. Post operatively Immobilization, Oral intake, Intravenous nutrition after study, Removal of nasogastric tube, Removal of catheter.

Intervention Abdominal drain group with ERAS protocol and no abdominal drain group with ERAS protocol.

Sample size calculation Sample size is calculated using "R". A sample size of 76 (38 per group) was calculated with the study powered at 90 percent, to prove that the no abdominal drain group is non inferior compared to the abdominal drain group in terms of length of hospital stay. The clinically relevant non inferiority margin was assumed is one day. The alpha error assumed 0.05 ( mention about loss to follow up. The pooled Standard deviation (SD) taken from previous study (done at our institute by Mishra TS et al) 1.5. Assuming a loss to follow up of 15 percent. The ultimate sample size was calculated to be 76+11=87. 87 cases will be taken on the whole to ensure equal distribution in both arms. Recruitment will be stopped at 76 cases along with necessary follow up or at 87 including loss to follow up which ever is achieved earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patient of peptic ulcer perforation peritonitis ( when confirmed intraoperatively)
* Perforation of size less than or equal to 1 cm.
* Patient age more than 18 years age
* American society of anesthesiologists score of I or II

Exclusion Criteria:

* Refractory septic shock at presentation
* Known Chronic kidney disease (CKD)/Chronic liver disease (CLD) patients
* Deranged LFT, RFT or active respiratory illness pneumonia or COPD ( Spo2 below 94 on room air)
* Pregnant patients
* History of chronic steroid abuse
* INTRAOPERATIVELY detected coexistent bleeding peptic ulcer, perforation requiring operation other than omental patch repair, spontaneously sealed peptic perforation, malignant perforation
* Patient requiring positive pressure ventilatory support post-operatively for more than 6 hours.
* Patient refusing consent.
* Co-existent neurological or psychiatric illness or unable to understand the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay (in days) | Post operative period up-to one month.
  Duration from the time of operation to time of discharge

SECONDARY OUTCOMES:
Early postoperative abdominal pain measured using the Verbal numeric scale (VNS) | At 8 hours, 24 hours and 72 hours postoperatively
  Verbal numeric scale (VNS) measured in the early postoperative period at different time frames as mentioned. Verbal numeric scale score will include score from 0 to10.On asking patient will grade his /her severity of pain between 0 to 10. 0 means the no pain and 10 means worst imaginable pain.
Time of recovery of Functional parameters (in hours) | Up to one month post operatively
  Onset of walk, onset of flatus, onset of stool, onset of liquid diet, onset of solid diet, onset of complete oral diet (discontinuation of IV fluids)
Incidence of Complications | Up-to one month post operatively
  Skin and soft tissue infection (SSI), Intra-abdominal Abscess, Abdominal wound dehiscence, Duodeno / gastro-cutaneous fistula, Post operative pneumonia, post operative paralytic ileus beyond 72 hours
Need for re-intervention in either arm | Up-to one month post operatively
  Number times an intervention is required for delay in recovery of functional parameters or an early complication e.g. reinsertion of Ryle's tube, Ultrasonography (USG) guided aspiration or drainage, or open drainage or re operation will be recorded
Re-admission rates | Date of discharge to 1 month post operative period
  Readmission for any post operative complications like fever/ or delayed functional recovery or any intervention will be recorded
Quality of life scoring and assessment | Post operative period - at 48 hours after surgery, at one month follow up and at third month follow up.
  Quality of life assessment will be done using EQ-5D-5L questionnaire (Euroqol 5 dimensions and 5 levels). It has 2 components, descriptive and objective. Descriptive component comprises of 5 dimensions which are mobility, self care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, namely no problem,0 slight problems, moderate problems, severe problems and extreme problems. Objective component is also called Euroqol visual analog scale. Score ranges from zero (the worst possible health status the participant can imagine) to 100 (the best possible health outcome the participant can imagine). It will be assessed on the day of discharge, follow up at one month and follow up at third month in the post operative period.
Degree of compliance to the ERAS protocol | Up to the time of discharge
  The degree of compliance to each of the parameters in the ERAS protocol will be recorded and expressed in percentage

CONTACTS AND LOCATIONS:
Overall Officials: TUSHAR S MISHRA, MBBS,MS,FACS, Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences,, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gonenc M, Dural AC, Celik F, Akarsu C, Kocatas A, Kalayci MU, Dogan Y, Alis H. Enhanced postoperative recovery pathways in emergency surgery: a randomised controlled clinical trial. Am J Surg. 2014 Jun;207(6):807-14. doi: 10.1016/j.amjsurg.2013.07.025. Epub 2013 Oct 10. PMID 24119887
- [Result] Mohsina S, Shanmugam D, Sureshkumar S, Kundra P, Mahalakshmy T, Kate V. Adapted ERAS Pathway vs. Standard Care in Patients with Perforated Duodenal Ulcer-a Randomized Controlled Trial. J Gastrointest Surg. 2018 Jan;22(1):107-116. doi: 10.1007/s11605-017-3474-2. Epub 2017 Jun 26. PMID 28653239
- [Result] Lohsiriwat V, Jitmungngan R. Enhanced recovery after surgery in emergency colorectal surgery: Review of literature and current practices. World J Gastrointest Surg. 2019 Feb 27;11(2):41-52. doi: 10.4240/wjgs.v11.i2.41. PMID 30842811
- [Result] Agarwal A, Jain S, Meena LN, Jain SA, Agarwal L. Validation of Boey's score in predicting morbidity and mortality in peptic perforation peritonitis in Northwestern India. Trop Gastroenterol. 2015 Oct-Dec;36(4):256-60. doi: 10.7869/tg.300. PMID 27509704